CLINICAL TRIAL: NCT05392946
Title: Phase 1/2 Trial of Iberdomide in Combination With Daratumumab, BortEzomib and DexamethAsone in Patients With Newly Diagnosed Multiple MyeLoma (IDEAL)
Brief Title: Iberdomide, Daratumumab, Bortezomib, and Dexamethasone for Treatment of Newly Diagnosed Multiple Myeloma, IDEAL Study
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC200807; NCI-2022-02414 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-006604 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-05-19; First posted 2022-05-26 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (iberdomide, bortezomib, dexamethasone, daratumumab) (Experimental): INDUCTION PHASE: Patients receive iberdomide PO QD on days 1-21, bortezomib SC on days, 1, 8, 15, and 22, and dexamethasone PO on days 1, 8, 15, 22. Patients also receive daratumumab SC on days 1, 8, 15, 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  CYCLES 13-36 CYCLES: Patients receive iberdomide PO QD on days 1-21. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Daratumumab; Drug: Dexamethasone; Drug: Iberdomide

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Biological: Daratumumab — Given SC
  Other Names: Darzalex; HuMax-CD38; JNJ-54767414; Daratumumab Biosimilar HLX15; Daratumumab-fihj
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Iberdomide — Given PO
  Other Names: CC 220; CC-220

SUMMARY:
This phase I/II trial studies the side effects and best dose of iberdomide and how well it works in combination with daratumumab, bortezomib, and dexamethasone in treating patients with newly diagnosed multiple myeloma. Immunotherapy with iberdomide, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Daratumumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving iberdomide in combination with daratumumab, bortezomib, and dexamethasone may kill more cancer cells in patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the maximum tolerated dose (MTD) of iberdomide in combination with daratumumab, bortezomib, and dexamethasone. (Phase 1 [Dose Confirmation Cohort]) II. To determine the complete response rate as best response during induction therapy with (1) iberdomide, daratumumab, bortezomib and dexamethasone (IberDVd) when used as initial therapy in patients with previously untreated symptomatic multiple myeloma. (Phase 2)

SECONDARY OBJECTIVES:

I. To assess the expanded response definition, overall response rate (ORR), and very good partial response (VGPR) rate of iberdomide in combination with daratumumab, bortezomib and dexamethasone. (Phase 2) II. To assess the progression free survival and overall survival among patients with previously untreated symptomatic multiple myeloma following treatment with iberdomide in combination with daratumumab, bortezomib and dexamethasone. (Phase 2) III. To assess the time to response (defined as the time between the date of first dose and the first documented evidence of a partial response or better) following treatment with iberdomide in combination with daratumumab, bortezomib and dexamethasone in patients with previously untreated symptomatic multiple myeloma (MM). (Phase 2) IV. To describe the toxicities associated with iberdomide in combination with daratumumab, bortezomib and dexamethasone in patients with previously untreated symptomatic MM and toxicities associated with dose attenuated iberdomide monotherapy administered from cycles 13 through 36. (Phase 2)

CORRELATIVE RESEARCH OBJECTIVES:

I. Examine the proportion of next generation flow cytometry assessed measurable residual disease (MRD) negative complete response following induction therapy with the combination of iberdomide in combination with daratumumab, bortezomib and dexamethasone. (Phase 2) II. To identify the proportion of patients with MRD negative complete response (as measured by the next-generation flow cytometry, sensitivity 10-5) at the end of cycles 24 and 36 during the deescalated phase of iberdomide monotherapy administration. (Phase 2) III. Examine the proportion of sustained MRD negative complete response following 6 months after attaining complete response (CR) and at the end of cycles 24 and 36. (Phase 2) IV. Evaluate pharmacokinetics and pharmacodynamics of iberdomide in combination with daratumumab, bortezomib and dexamethasone. (Phase 2)

OUTLINE: This is a phase I, dose-escalation study of iberdomide followed by a phase II study.

INDUCTION PHASE: Patients receive iberdomide orally (PO) once daily (QD) on days 1-21, bortezomib subcutaneously (SC) on days, 1, 8, 15, and 22, and dexamethasone PO on days 1, 8, 15, 22. Patients also receive daratumumab SC on days 1, 8, 15, 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

CYCLES 13-36 CYCLES: Patients receive iberdomide PO QD on days 1-21. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.

Patients also undergo bone marrow aspiration and/or biopsy, magnetic resonance imaging (MRI) or positron emission tomography (PET) and computed tomography (CT) scan, and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at the time of signing the informed consent form (ICF)
* Previously untreated active/symptomatic multiple myeloma or have received no more than one cycle of any anti-myeloma treatment regimen for active/symptomatic myeloma

  * NOTE: Prior radiation therapy for the treatment of solitary plasmacytoma is permitted. Prior therapy with clarithromycin, dehydroepiandrosterone (DHEA), anakinra, pamidronate or zoledronic acid is permitted. Any additional agents not listed must be approved by the principal investigator
* Measurable disease

  * Serum M-protein ≥0.5 g/dL
  * Urine M-protein ≥200 mg in a 24-hour collection
  * Serum Free Light Chain level ≥ 10 mg/dL provided the free light chain ratio is abnormal
  * Measurable plasmacytoma [at least one lesion that has a single diameter of ≥2 cm on positron emission tomography (PET)-computed tomography (CT) scan]
  * Bone marrow plasma cells≥30%
  * Patients with IgA myeloma in whom serum protein electrophoresis is deemed unreliable, due to co-migration of normal serum proteins with the para protein in the beta region, may be considered eligible as long as total serum IgA level is elevated above normal range.
  * For patients with extramedullary disease (EMD) measurable by CT or MRI or the CT portion of the PET/CT: Must have at least one lesion that has a single diameter of ≥2 cm. Skin lesions can be used if the area is ≥2cm in at least one diameter and measured with a ruler.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Hemoglobin >= 8.0 g/dL (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (Exception for Gilbert's syndrome) (obtained =< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 2 x ULN and alkaline phosphatase =< 1.5 x ULN (obtained =< 14 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy (obtained =< 14 days prior to registration)
* Calculated creatinine clearance >= 50 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only. Note: A person of childbearing potential (PCBP) is a person who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) and must:

  * Have 2 negative pregnancy tests as verified by the Investigator prior to starting study treatment and must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact. AND
  * Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with two forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting investigational product, during the study treatment, and for at least 28 days after the last dose of Iberdomide (90 days after the last dose of daratumumab, 7 months after last dose of bortezomib whichever is longer).
  * NOTE: Non-childbearing potential is defined as follows (by other than medical reasons):

    * >= 45 years of age and has not had menses for > 24 months
    * Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
    * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure
* Willingness to follow Pregnancy Prevention Program requirements:

  * Persons of childbearing potential must agree to use a contraceptive method that is highly effective (with a failure rate of < 1% per year), preferably with low user dependency, during the intervention period and for at least 7 months after the last dose of study intervention. These patients must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period
  * Persons able to father a child must agree that during the treatment intervention period and for 6 months after the last dose of study treatment (to allow for clearance of any altered sperm), the participant will:

    * Refrain from donating sperm while on study treatment, during dose interruptions and for at least 6 months following last dose of study treatment, PLUS either:

      * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR,
      * Must agree to use contraception/barrier such as a male condom (even if they have undergone successful vasectomy), and when having sexual intercourse with a person of childbearing potential who is not currently pregnant his partner will use an additional highly effective contraceptive method with a failure rate of < 1% per year
* Provide written informed consent
* Negative hepatitis B test (defined by a negative test for hepatitis B surface antigen [HBsAg], or antibodies to hepatitis B surface and/or core antigens [antiHBs or antiHBc)

  * NOTE: Participants with resolved hepatitis B infection (i.e.., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded from the study.
  * NOTE: Participants with serologic findings suggestive of hepatitis B virus (HBV) vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior HBV vaccination do not need to be tested for HBV deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR). Those who are PCR positive will be excluded from the study
* Willingness to provide mandatory bone marrow specimens for correlative research
* Willing and able to adhere to the study visit schedule and other protocol requirements. Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willing to refrain from donating blood while on study treatment, during dose interruptions and for at least 28 days following the last dose of study treatment

Exclusion Criteria:

* Monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, or AL amyloidosis
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Receiving any other concurrent chemotherapy, or any ancillary therapy considered investigational

  * NOTE: Bisphosphonates are considered to be supportive care rather than therapy and are thus allowed while on protocol treatment
* Known to be human immunodeficiency virus (HIV) positive, known or suspected active hepatitis C infection or seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]) at screening or within 3 months prior to first dose of study treatment.

  * NOTE: Participants with resolved hepatitis B infection (i.e.., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded.
  * EXCEPTION: subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection (defined as infection undergoing treatment)
  * Active mucosal or internal bleeding,
  * Social situations that would limit compliance with study requirements (including drug addiction)
  * Known gastrointestinal disease (including difficulty swallowing) or gastrointestinal procedure that could interfere with the oral absorption or tolerance of iberdomide or dexamethasone
  * Unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. NOTE: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria
  * Active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). NOTE: Participants with isolated proteinuria resulting from MM are eligible, provided they fulfil inclusion criteria
* Evidence of cardiovascular disease risk, as defined by any of the following:

  * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block
  * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three (3) months of Screening
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system
  * Uncontrolled hypertension
  * History of life-threatening ventricular arrhythmias
* Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) 50% of predicted normal. Note that forced expiratory testing (FEV1) is required for subjects suspected of having COPD and subjects must be excluded if FEV1 is < 50% of predicted normal
* Known moderate or severe persistent asthma, or currently has uncontrolled asthma of any classification
* Acute diffuse infiltrative pulmonary and pericardial disease
* Unable or unwilling to undergo protocol required thromboembolism prophylaxis
* Has taken a strong inhibitor or inducer of CYP3A4/5 including grapefruit, St. John's Wort or related products =< 14 days prior to registration
* Known allergy to any of the study medications, their analogues or excipients in the various formulations
* Major surgery =< 14 days prior to registration
* Plasmapheresis =< 14 days prior to registration
* Has been treated with an investigational agent (i.e., an agent not commercially available) =< 28 days or 5 half-lives (whichever is longer) prior to registration
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Radiotherapy =< 14 days prior to registration

  * NOTE: If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the iberdomide
* More than 1 prior cycle of an antimyeloma therapy or corticosteroids for the treatment of active / symptomatic multiple myeloma by SLiMCRAB criteria

  * NOTE: Prior corticosteroid use for the treatment of non-malignant disorders is permitted
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Peripheral neuropathy >= grade 3 on clinical examination or grade 2 with pain during the screening period
* Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L)
* Gastrointestinal disease that may significantly alter the absorption of iberdomide
* History of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, pomalidomide, or pegfilgrastim / biosimilars
* The subject has a planned or received immunization with a live or live attenuated vaccine =< 8 weeks prior to registration
* History of prior malignancies, other than MM, unless the subject has been free of the disease for >= 5 years with the exception of the following noninvasive malignancies:

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast
  * Incidental histological findings of prostate cancer such as T1a or T1b using the Tumor/Node/Metastasis (TNM) classification of malignant tumors or prostate cancer that is curative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of iberdomide (Phase I) | Up to 12 cycles. Each cycle is 28 days.
  MTD is defined as the highest tested dose level that is determined to have acceptable toxicity and tolerability based on dose limiting toxicity definitions.
Complete response rate (Phase II) | Up to 3 years
  A confirmed complete response is defined as a patient who has achieved an stringent complete response (sCR) or complete response (CR) and maintained it on two consecutive evaluations at any time during induction therapy. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. 95% confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Overall response rate (Phase II) | Up to 3 years
  Will be estimated by the total number of patients who achieve a sCR, CR, very good partial response (VGPR), or partial response divided by the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
VGPR or better response rate (Phase II) | Up to 3 years
  Will be estimated by the total number of patients who achieve at least a VGPR divided by the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true VGPR or better response rate will be calculated.
Progression-free survival (Phase II) | Up to 3 years
  Assessed as the time from registration to the earliest date of documentation of disease progression or death due to any cause. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Overall survival (Phase II) | Up to 3 years
  Assessed as from registration to death due to any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Incidence of adverse events (AEs) (Phase II) | Up to 30 days after discontinuation
  The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns.
Proportion of patients with measurable residual disease (MRD) negative complete response (Phase II) | At the end of cycles 24 and 36. Each cycle is 28 days
  The proportion of patients who achieve MRD negative complete response at the end of cycles 24 and 36 will be estimated by the number of patients who are MRD negative (as measured by the next-generation flow cytometry, sensitivity 10-5) at the end of end of cycles 24 and 36 divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true MRD negative rates end of cycles 24 and 36 of therapy will be calculated.

OTHER OUTCOMES:
Minimal residual disease | Up to 3 years
  Will be assessed on bone marrow aspirate in all patients achieving sCR or CR. The proportion of patients who achieve MRD negative status following induction will be estimated by the number of patients who are MRD negative at the end of induction divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true MRD negative rate after induction will be calculated.
Proportion of patients who achieve sustained MRD negative status | At the end of cycles 24 and 36. Each cycle is 28 days.
  Will be estimated by the number of patients who are MRD negative at the end of end of cycles 24 and 36 divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true MRD negative rates end of cycles 24 and 36 of therapy will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kapoor, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials